Official Title: The Effects of Electrical Muscle Stimulation Exercise on Upper, Lower

Extremity and Core Strength in Sedentary Women

NCT Number: Pending

Date: October 7, 2025

Prepared by: Dr. Ali Kerim Yılmaz

Esra Korkmaz Salkılıç

Institution: 19 Mayıs University

## The Effect of Electrical Muscle Stimulation Exercise on Lower, Upper Extremity, and Core Strength in Sedentary Women

## **Statistical Analysis**

SPSS 21.0 package program was used for data analysis. The normality assumption of the data was examined with the Kolmogorov-Simirnov test and it was determined that the variables were normally distributed (p>0.05). One-way analysis of variance in repeated measures and Mixed Design Analysis of Variance in Repeated Measures were applied to the data. Sphericity was examined with Mauchly's Sphericity test. The Sphericity Assumed test was used for those with equal variances (p>0.05). In cases where variances were not equal (p<0.05), the epsilon value ( $\epsilon$ ) was examined and Greenhouse and Geisser tests were used when  $\epsilon$ 0.75 and Huynh-Feldt tests were used when  $\epsilon$ 0.75. Bonferroni test was used to determine the intergroup differences. Data were presented as mean and standard deviation and evaluated at a significance level of p<0.05.